CLINICAL TRIAL: NCT05675267
Title: Interest of the HEART Score for the Management of Patients With Chest Pain in Emergency Department
Acronym: HEART-SAU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_019_HEART-SAU
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; chest pain; emergency department; HEART score
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with chest pain
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — HEART score calculation

SUMMARY:
Chest pain is a frequent reason of consultation in emergency department. Emergency physician have to identify patients at high risk of Acute Coronary Syndrome from those presenting a lower risk.

DETAILED DESCRIPTION:
The aim of the study is to study the interest of the HEART score for the management of patients with chest pain in emergency department

ELIGIBILITY:
Inclusion Criteria:

men and women Aged more than 18 Chest pain Consulting in emergency department Agreeing to participate to the study

Exclusion Criteria:

aged less than 18 not agreeing to participate to the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient with chest pain consulting in emergency department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
HEART score | Day 0
  Cardiovascular risk evaluated using HEART score. HEART score includes 5 items on history of chest pain, electrocardiogram, patient's age, cardiovascular risk factors and initial troponin. Each item is coded from 0 to 2 points, the overall score ranges from 0 to 10 points. Score between 0 and 3 indicated low risk of major adverse cardiovascular event, Score between 4 and 6 indicated moderate risk of major adverse cardiovascular event, Score between 7 and 10 indicated high risk of major adverse cardiovascular event